CLINICAL TRIAL: NCT00001184
Title: A Natural History Study of the Immune Regulation of Idiopathic Inflammatory Bowel Diseases: Crohn's Disease, Ulcerative Colitis, and Other Inflammatory Conditions of the Gut
Brief Title: Immune Regulation in Ulcerative Colitis or Crohn s Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 820183; 82-I-0183
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Chrohn's Disease
Keywords: CGD related IBD; IBD Hermansky-Pudlak Syndrom; Natural History
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients between the ages of 0 and 75 years of age with Crohn s disease or ulcerative colitis or symptoms of inflammatory bowel disease may be eligible for this study.

SUMMARY:
This study will investigate in patients with Crohn s disease and ulcerative colitis how the body s immune system controls inflammation in the gastrointestinal tract (stomach and intestines)-specifically, how lymphocytes (a type of white blood cell) function in inflammatory responses. This protocol does not involve any experimental treatments.

Patients between the ages of 0 and 75 years of age with Crohn s disease or ulcerative colitis or symptoms of inflammatory bowel disease may be eligible for this study. Screening tests may include the following: medical history and physical examination, routine blood tests, examination of stool specimens, X-rays such as barium enema or upper GI series, proctosigmoidoscopy, colonoscopy, gastroduodenoscopy, and small bowel biopsy.

Participants will receive medical treatment according to the best generally accepted measures for treating Crohn s disease or ulcerative colitis. This may include anti-inflammatory drugs, immunosuppressive drugs, and antibiotics to treat infections. A surgical consultation may be recommended for patients whose disease does not respond to medical treatment. If surgery to remove intestinal tissue is recommended, a qualified gastrointestinal surgeon will perform the procedure.

In addition, participants may undergo the following procedures:

* Blood drawing - No more than 450 milliliters (30 tablespoons, or 15 ounces) of blood will be taken from adults over a 6-week period. A maximum of 7 ml (1/2 tablespoon) of blood per kilogram (2.2. pounds) of body weight will be obtained from children within the same time period, with no more than 3 ml/kg taken at any one time.
* Leukapheresis - This procedure is done to collect large quantities of white blood cells. Whole blood is collected through a needle in an arm vein, similar to donating blood. The blood is circulated through a machine that separates it into its components, and the white cells are removed. The rest of the blood is returned to the body, either through the same needle or through another needle in the other arm.
* Intestinal biopsies - Intestinal tissue will be obtained during colonoscopy with intestinal biopsy in patients who require this procedure as part of their standard medical care. Patients are given a sedative to reduce anxiety, but are conscious during the procedure. A flexible tube is inserted into the rectum and large intestine, allowing the physician to see the intestinal mucosa. At various places, small pieces of tissue are plucked out.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

This natural history protocol provides for the evaluation of patients with idiopathic inflammatory bowel diseases (ulcerative colitis, Crohn s disease, IBD associated with immunodeficiency and genetic diseases such as chronic granulomatous disease, and additional undefined inflammatory conditions of the gut) either on an inpatient or outpatient basis.

OBJECTIVES:

Primary Objective: To identify the molecular abnormalities that result in inflammatory bowel diseases and develop novel therapies based on these discoveries.

Secondary Objectives: To enroll patients with IBD in order to obtain clinical, therapeutic, immunological, and genetic data relevant to the research study of their disease.

ENDPOINTS:

Primary Endpoint: Comparison of the molecular and cellular abnormalities that result in inflammatory bowel diseases

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients with a verifiable diagnosis of Crohn s disease, ulcerative colitis, or IBD known to be associated with a co-existing condition and which is supported by characteristic clinical features, radiographic or endoscopic findings, or consistent histopathologic mucosal

     changes OR
  2. Patients with clinical features consistent with an unclassified inflammatory bowel disease and histologic evidence of inflammation of the intestine OR
  3. Patients with any clinical features consistent with inflammatory bowel disease (intestinal inflammation), including but not limited to abdominal pain, fistulae, weight loss, diarrhea, hematochezia or melena or suggestive extra-intestinal symptoms (pyoderma, erythema

     nodosum, axial and articular arthralgias, uveitis, fatigue, fever), in which a diagnosis has not been verified. OR
  4. Patients who have a defined genetic syndrome linked to inflammatory bowel disease risk with or without symptoms or findings consistent with IBD
  5. All subjects to be enrolled will be between ages 0-75 (Participants coming to the NIH Clinical Center must meet age and weight requirements of the clinical center, but > 18 must years old for patients without IBD and may be as young as 0-2 years old for mail-in

     samples).
  6. To participate in the research biopsies during endoscopy, subjects must have the following lab values within two weeks of the procedure:

     * Hematocrit > 30%
     * Platelet count > 100,000
     * PT INR < 1.3 or PTT prolonged by < 3 seconds
  7. Ability to consent to the protocol on their own.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

1. Must be willing to undergo blood draw and/or upper endoscopy and colonoscopy with biopsy to obtain material for research purposes.
2. Must be >=18 years old.
3. Must be willing to submit samples for storage.

INCLUSION OF EMPLOYEES IN THE NIH INTRAMURAL STUDIES:

NIH employees and members of their immediate families may participate in this protocol. We will follow the Guidelines for the Inclusion of Employees in NIH Research Studies and will give each employee a copy of the NIH information sheet on Employee Research Participation.

For NIH employees:

1. Neither participation nor refusal to participate will have an effect, either beneficial or adverse, on the participant s employment or work situation.
2. The NIH information sheet regarding NIH employee research participation will be distributed to all potential subjects who are NIH employees.
3. The employee subject s privacy and confidentiality will be preserved in accordance with NIH Clinical Center and NIAID policies, which define the scope and limitations of the protections.
4. For NIH employee subjects, consent will be obtained by an individual independent of the employee s team. Those in a supervisory position to any employee and co-workers of the employee will not obtain consent. The protocol study staff will be trained annually on obtaining potentially sensitive and private information from co-workers or subordinates. This training will be reinforced as needed, at weekly team meetings.

EXCLUSION CRITERIA:

1. Failure to meet the inclusion criteria.
2. Any medical, psychiatric, or social conditions which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the subject.

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

1. History of inflammatory bowel disease.
2. Acute systemic or intestinal infection requiring antibiotics
3. Any condition that, in the investigator s opinion, places the patient at undue risk by participating in the study.

Ages: 1 Day to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinical
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 1998-08-07 (Actual)

PRIMARY OUTCOMES:
To identify the molecular abnormalities that result in inflammatory bowel diseases and develop novel therapies based on these discoveries. | at close of study
  observational

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Fuss, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1982-I-0183.html